CLINICAL TRIAL: NCT01807728
Title: Training Programs to Improve Outcomes for Individuals With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Boninger, Chair, Department of Physical Medicine and Rehabilitation, University of Pittsburgh
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 12090536; H133A120004 (Other Grant/Funding Number: U.S. Department of Education)
Record Dates: First submitted 2013-03-01; First posted 2013-03-08 (Estimated); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Spinal Cord Injuries
Keywords: Quality of life; Participation; Training
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 Training Program (Experimental): For Group 1, participants will aim to be recruited within the first week of their inpatient rehabilitation stay (admission time point).
  Interventions: Other: Group 1 Training Program
- Group 2 Training Program (Experimental): For Group 2, individuals may be enrolled in the study at any time over their inpatient rehabilitation stay. Data collection may occur at admission (Group 2 only), just prior to discharge and at 3, 6 and 12 months after discharge.
  Interventions: Other: Group 2 Training Program

INTERVENTIONS:
Other: Group 1 Training Program — Up to four group classes which will involve peer interaction, hands on training activities, and interaction with group leader(s).
  Arms: Group 1 Training Program
Other: Group 2 Training Program — Two group classes which will involve peer interaction, hands on training activities, and interaction with group leader(s).
  Arms: Group 2 Training Program

SUMMARY:
The objective of this study is to determine the effectiveness of different training programs on outcomes in persons with spinal cord injury (SCI). We are interested to see which programs have the greatest impact.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years old
* Use either a power or manual wheelchair as a primary means of mobility (>50% of weekly mobility)
* Living in the community
* Must have a non-progressive spinal cord injury
* Manual wheelchair users must be able to independently propel their wheelchairs
* Manual wheelchair users score ≤90 on the Wheelchair Skills Training Questionnaire (WST-Q)

Exclusion Criteria:

* Cognitive impairment that could interfere with learning

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2018-03-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in quality of life at 1 year | Baseline, 1 Year
  Predict mode of mobility at 1 year post-discharge based on patient characteristics and activity during IPR using a minimum data collection window. Predict ambulatory ability at 1 year post-discharge based on patient characteristics and measures of non-purposeful activity.

SECONDARY OUTCOMES:
Change from baseline in quality of life at 1 month | Baseline, 1 month
  Predict mode of mobility at discharge or 1 month based on patient characteristics and activity during IPR using a minimum data collection window. Predict ambulatory ability at discharge or 1 month based on patient characteristics and measures of non-purposeful activity.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Boninger, MD, Principal Investigator — University of Pittsburgh
Locations (4):
- United States (4):
  - South Florida Spinal Cord Injury System, Miami, Florida
  - Midwest Regional Spinal Cord Injury Care System, Chicago, Illinois
  - Northern New Jersey Spinal Cord System, West Orange, New Jersey
  - Debbie, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Worobey LA, McKernan G, Toro M, Pearlman J, Cowan RE, Heinemann AW, Dyson-Hudson TA, Pedersen JP, Mesoros M, Boninger ML. Effectiveness of Group Wheelchair Maintenance Training for People with Spinal Cord Injury: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2022 Apr;103(4):790-797. doi: 10.1016/j.apmr.2021.02.031. Epub 2021 Jun 24. PMID 34174224
- [Derived] Worobey LA, Kirby RL, Cowan RE, Dyson-Hudson TA, Shea M, Heinemann AW, Pedersen JP, Hibbs R, Boninger ML. Using remote learning to teach clinicians manual wheelchair skills: a cohort study with pre- vs post-training comparisons. Disabil Rehabil Assist Technol. 2022 Oct;17(7):752-759. doi: 10.1080/17483107.2020.1804633. Epub 2020 Aug 18. PMID 32809896